CLINICAL TRIAL: NCT01301131
Title: Randomized Controlled Trial of Fermented Dairy Product Containing L. Casei Shirota for Prevention of Ventilator-Associated Pneumonia
Brief Title: Probiotics for Prevention of Ventilator-Associated Pneumonia (VAP)
Acronym: VAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Visanu Thamlikitkul, Faculty of Medicine Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SirirajCEU 54-002
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Drug Safety
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental): 80 ml of fermented dairy product containing L. casei shirota via nasogastric tube once daily and 80 ml of fermented dairy product containing L. casei shirota oral rinse once daily
  Interventions: Other: Probiotics
- control (No Intervention)
  Interventions: Other: control

INTERVENTIONS:
Other: Probiotics — 80 ml of fermented dairy product containing L. casei shirota via nasogastric tube once daily and 80 ml of fermented dairy product containing L. casei shirota oral rinse once daily
  Other Names: Yakult
  Arms: Probiotic
Other: control — usual oral care
  Other Names: regular care
  Arms: control

SUMMARY:
Hospitalized patients with ventilator are randomized to receive fermented dairy product containing L. casei shirota or nothing. The main outcome is development of ventilator-associated pneumonia (VAP)

DETAILED DESCRIPTION:
Fermented dairy product containing L. casei shirota has bee shown to inhibit multi-drug-resistant bacteria. This study is conducted to determine if Fermented dairy product containing L. casei shirota can prevent ventilator-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

Patient age ≥ 18-year who received ventilator and agreed to participate by signing informed consent form

Exclusion Criteria:

Immunocompromised host (e.g. HIV infection, On immunosupressive agents, ANC ≤ 500 cell/ml), Pregnancy, History of congenital heart disease, rheumatic fever, previously infective endocarditis, prosthetic valve, Contraindication for enteral feeding, History of milk or milk-product allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with pneumonia | up to 28 days
  patient with pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Visanu Thamlikitkul, MD, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand